CLINICAL TRIAL: NCT05295589
Title: A Randomized Phase II Trial Comparing the Combination of PI3K Inhibitor Copanlisib (BAY 80-6946) and PARP Inhibitor Olaparib (AZD2281) to Standard Chemotherapy in Patients With Recurrent Platinum Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Have Progressed Through Prior PARP Inhibitor Therapy
Brief Title: Comparing Standard of Care Chemotherapy Treatment to the Combination of Copanlisib and Olaparib for Recurrent Platinum Resistant Ovarian Cancer That Has Progressed Through PARP Inhibitor Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-02228; NCI-2022-02228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY029 (Other: NRG Oncology); NRG-GY029 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-03-23; First posted 2022-03-25 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Platinum-Refractory Fallopian Tube Carcinoma; Platinum-Refractory Ovarian Carcinoma; Platinum-Refractory Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Endometrioid Adenocarcinoma; Recurrent Fallopian Tube High Grade Serous Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian High Grade Serous Adenocarcinoma; Recurrent Platinum-Resistant Fallopian Tube Carcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma; Recurrent Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Endometrioid Adenocarcinoma; Recurrent Primary Peritoneal High Grade Serous Adenocarcinoma
MeSH Terms: interventions — copanlisib; Magnetic Resonance Spectroscopy; olaparib; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care chemotherapy) (Active Comparator): Patients receive either paclitaxel IV OR pegylated liposomal doxorubicin hydrochloride IV, OR topotecan hydrochloride IV while on study.
  Patients undergo CT scan while on study and may undergo MRI throughout the study.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Topotecan Hydrochloride
- Arm II (copanlisib, olaparib) (Experimental): Patients receive copanlisib hydrochloride IV and olaparib PO while on study. Patients undergo CT scan while on study and may undergo MRI throughout the study.
  Interventions: Procedure: Computed Tomography; Drug: Copanlisib Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Olaparib

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Copanlisib Hydrochloride — Given IV
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
  Arms: Arm II (copanlisib, olaparib)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
  Arms: Arm II (copanlisib, olaparib)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (standard of care chemotherapy)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm I (standard of care chemotherapy)
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm I (standard of care chemotherapy)

SUMMARY:
This phase II trial compares copanlisib and olaparib to standard of care chemotherapy in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that did not respond to previous platinum-based chemotherapy (platinum resistant) and that has come back (recurrent). Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Olaparib is a PARP inhibitor. PARP is a protein that helps repair damaged deoxyribonucleic acid (DNA). Blocking PARP may prevent tumor cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving copanlisib and olaparib may extend the time that the cancer does not progress compared to standard of care chemotherapy in patients with recurrent platinum resistant ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the clinical efficacy of the combination of copanlisib/olaparib, as measured by investigator-assessed progression free survival (PFS), compared to standard chemotherapy in the setting of recurrent platinum resistant ovarian cancer that has progressed through prior PARP inhibitor therapy.

SECONDARY OBJECTIVES:

I. To assess the clinical efficacy of the combination of copanlisib/olaparib, as measured by objective response rate (ORR), per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To assess the clinical efficacy of the combination of copanlisib/olaparib, as measured by overall survival (OS), compared to standard chemotherapy in the setting of recurrent platinum resistant ovarian cancer that has progressed through prior PARP inhibitor therapy.

III. To determine the nature, frequency and degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5.0 for each treatment arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive either paclitaxel intravenously (IV) OR pegylated liposomal doxorubicin hydrochloride IV, OR topotecan hydrochloride IV while on study.

ARM II: Patients receive copanlisib hydrochloride IV and olaparib orally (PO) while on study.

Patients undergo computed tomography (CT) scan while on study and may undergo magnetic resonance imaging (MRI) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent ovarian cancer. Ovarian cancer = fallopian tube cancer, ovarian cancer, primary peritoneal cancer. The following histology types are eligible:

  * High grade serous
  * Endometrioid, grade 3
  * Any histology with BRCA1 and/or BRCA2 deleterious mutation (germline or somatic)

    * Histologic confirmation of the original primary tumor is required via the pathology report (upload of report required)
    * Confirmation of BRCA1 and BRCA2 germline status is required for all entered patients (upload of report[s] required)
    * Tumor/somatic genomic testing can be provided or entered as not done (upload of report[s] required)
    * Homologous recombination deficiency (HRD) testing can be provided or entered as not done (upload of report[s] required)
    * Genetic/genomic testing results and HRD testing results, initially entered as not done, should be uploaded if they become available anytime during conduct of the study
* Participants must have progressed by imaging while receiving PARP inhibitor therapy (irrespective of whether PARP inhibitor therapy was given as maintenance therapy or as primary recurrence therapy); rising CA125 only is not considered as evidence of progression
* Platinum-resistant disease, defined as progression within < 6 months from completion of platinum-based therapy, and inclusive of platinum refractory disease. The date should be calculated from the last administered dose of platinum therapy
* Unlimited lines of cytotoxic therapy allowed in the platinum-sensitive setting; =< 2 lines of cytotoxic therapy allowed in the platinum-resistant setting

  * Hormonal therapy (e.g., tamoxifen, aromatase inhibitors) will not count as a previous line of therapy
* Prior use of bevacizumab in the upfront or recurrent setting is required
* Participants must have evaluable disease - defined as RECIST 1.1 measurable disease OR non-measurable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related in the setting of a CA125 > 2 x upper limit of normal [ULN])
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or 2
* Absolute neutrophil count (ANC) >= 1,500/mcl (within 14 days prior to registration)
* Hemoglobin >= 10 g/dL (within 14 days prior to registration)
* Platelets >= 100,000/mcL (within 14 days prior to registration)
* Creatinine clearance (CrCL) >= 51 mL/min (estimated using Cockcroft-Gault equation) (within 14 days prior to registration)
* Total serum bilirubin level =< 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (within 14 days prior to registration)
* Lipase =< 1.5 x ULN within 14 days of registration
* International normalized ratio (INR) =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 times the upper limit of normal within 14 days of registration
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional classification. To be eligible for this trial, patients should be class 2B or better
* Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose and INR/PTT is stable. Oral anticoagulants are allowed provided there are no interactions
* The effects of copanlisib and olaparib on the developing human fetus are unknown. For this reason and because maternal toxicity, developmental toxicity and teratogenic effects have been observed in nonclinical studies and PI3K inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 1 month after the last dose of copanlisib and/or olaparib. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and must be off steroids and stable at least one month
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Prior therapy:

  * No chemotherapy or radiotherapy within 4 weeks of registration
  * No hormonal therapy within 2 weeks of registration. Patients receiving raloxifene for bone health as per Food and Drug Administration (FDA) indication may remain on raloxifene absent other drug interactions
  * No investigational agents within 4 weeks of registration
  * No prior PI3K-AKT-mTOR pathway inhibitor therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib, copanlisib, or other agents used in this study
* Copanlisib and olaparib are primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted from 14 days prior to registration until the end of the study
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study. Patients may be using topical or inhaled corticosteroids
* Use of concomitant herbal medications/preparations (except for vitamins), alternative/complimentary medications, immunosuppressive therapy, or other prohibited medications
* Patients with uncontrolled type I or II diabetes mellitus; uncontrolled diabetes is defined as glycosylated hemoglobin (HbAlc) > 8.5%
* Patients with arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 3 months before registration
* Gastrointestinal conditions that would preclude consumption (swallowing), retention, and/or absorption of oral medications
* Patients with drainage gastrostomy tube are not allowed
* Patients with dependency on IV hydration or total parenteral nutrition (TPN) are not allowed
* Patients with uncontrolled intercurrent illness, including but not limited to:

  * Persistent grade >= 2 adverse events due to prior anti-cancer therapy with the exception of alopecia, hypothyroidism requiring medication, vitiligo, and the laboratory values defined in the inclusion criteria.
  * Known psychiatric illness/social situations that would limit compliance with study requirements.
  * History of or current autoimmune disease
  * Non-healing wound, ulcer, or bone fracture
  * Active, clinically serious infections > grade 2 (CTCAE v5.0)
* Women who are pregnant or unwilling to discontinue nursing
* Patients who have a history of non-infectious pneumonitis/interstitial lung disease (ILD) that required steroids, or current non-infectious pneumonitis/ILD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-03-17 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Time from study entry to time of progression or death, whichever occurs first, assessed up to 5 years
  The interim and primary analyses of PFS will be based on a logrank test, stratified by the factors declared at randomization. These analyses will include all patients enrolled onto the study regardless of compliance to their assigned study regimen. Patients will be grouped by their randomized treatment for intention-to-treat analyses. For the purposes of the primary analyses, the documentation of disease progression will be determined by the treating physician. The treatment hazard ratios and their 95% confidence intervals will be estimated using a multivariable proportional hazards model specified with main effects for the randomized treatment assignment (Arm 2 versus [vs] Arm 1) and covariate adjustment for the stratification factors declared at randomization.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  Defined as the binomial proportion of evaluable patients with a best overall response of complete response (CR) or partial response (PR) (by Response Evaluation Criteria in Solid Tumors 1.1). Responses reported by the treating physician will be used for these analyses. The ORR estimates by treatment arm will be supported by their 2-sided, 95% Wilson-Score confidence intervals (Wilson, 1927, Agresti, 1998). The relative odds of response in the experimental group (vs. the reference group) will be estimated using a multivariable logistic regression model specified with main effects for the treatment group and covariate adjustments for the stratification factors reported at baseline.
Overall survival (OS) | Time from study entry to time of death or the date of last contact, assessed up to 5 years
  The OS treatment hypothesis test will be based on a logrank test, stratified by the factors specified at randomization. The treatment hazard ratios and their 95% confidence intervals will be estimated using a multivariable proportional hazards model specified with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and covariate adjustment for the stratification factors used in the randomization.
Incidence of adverse events | Up to 5 years
  The nature, frequency, and degree of toxicity will be tabulated at the System Organ Class and adverse event-specific term levels using Common Terminology Criteria for Adverse Events version 5.0. Each patient will be represented according to the maximum grade observed for each term. Tabulations will show the number and percentage of patients by maximum grade, within the treatment group received, regardless of the randomized treatment assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis A Konstantinopoulos, Principal Investigator — NRG Oncology
Locations (5):
- United States (5):
  - University of Colorado Hospital, Aurora, Colorado
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT05295589/Prot_SAP_000.pdf